CLINICAL TRIAL: NCT02228759
Title: Ambulatory Continuous Adductor Canal Block to Facilitate Same Day Discharge Following Total Knee Arthroplasty: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Sugantha Ganapathy, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 105097
Record Dates: First submitted 2014-08-18; First posted 2014-08-29 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Knee Osteoarthritis
Keywords: Ambulatory home regional; adductor canal block; Postoperative pain; total knee arthroplasty; Home regional; Fast track arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee; Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adductor canal block (Experimental): The study is an open label pilot study to determine the feasibility of same day discharge following total knee arthroplasty with the use of a fast track regimen employing motor sparing knee blocks. The study will be performed on 25 American Society of Anesthesiologists class (ASA) 1-2 patients satisfying the inclusion criteria and undergoing unilateral primary total knee arthroplasty. First and second patients of the day undergoing surgery between Monday to Thursday in a week will be accessed for the study.
  Interventions: Procedure: Adductor canal block

INTERVENTIONS:
Procedure: Adductor canal block — All patients will recieve fast tracking with reduced fasting times, multimodal analgesia and adductor canal block

SUMMARY:
Patients scheduled to undergo total knee arthroplasty will receive motor sparing knee blocks with continuous adductor canal block along with multimodal analgesia started pre-operatively and continued into the postoperative period. The study will evaluate the feasibility of home discharge within the first 24 hours following total knee arthroplasty. We will also evaluate the pain scores in the first 5 days following the surgery, causes of delayed discharge and any adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Male and females of 40-70years of age
2. Scheduled to undergo unilateral primary total knee arthroplasty
3. ASA Class I, II

Exclusion Criteria:

1. ASA 3, 4
2. Revision surgery
3. Narcotic dependent (opioid intake morphine equivalent > 10 mg/ day for more than 3 months)
4. Other sources of chronic pain like fibromyalgia
5. Patients with associated significant cardiac, CNS or respiratory disease (poor cardio-respiratory reserve)
6. Major conduction defects in EKG (bifascilular block, CHB); significant valvular heart disease
7. Recent MI/ Stroke/ CHF (in the past 3 months)
8. BMI> 35
9. Obstructive sleep apnea (AHI > 15)
10. Patients with coexisting hematological disorder or with deranged coagulation parameters.
11. Patients with pre-existing major organ dysfunction such as hepatic and renal failure.
12. Psychiatric illnesses
13. Uncontrolled diabetes mellitus
14. Lack of informed consent.
15. Allergy to any of the drugs used in the study
16. Preoperative neurological deficits
17. Use of walking aids preoperatively
18. Living alone (Lack of Chaperone/home help)
19. Language barrier
20. Contralateral leg weakness
21. Pregnancy

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
percentage of patients discharged at 23 hours based on a composite of various factors represented on a pre-determined criteria | 24 hours

SECONDARY OUTCOMES:
first 24 hour pain scores | 24 hours
first 96 hour pain scores | 96 hours
Rescue analgesic frequency | 24 hours
total analgesic usage in the first 24 and 96 postoperative hours | 96 hours

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital, London Health Sciences centre, London, Ontario, Canada

REFERENCES:
- [Background] Ilfeld BM, Le LT, Meyer RS, Mariano ER, Vandenborne K, Duncan PW, Sessler DI, Enneking FK, Shuster JJ, Theriaque DW, Berry LF, Spadoni EH, Gearen PF. Ambulatory continuous femoral nerve blocks decrease time to discharge readiness after tricompartment total knee arthroplasty: a randomized, triple-masked, placebo-controlled study. Anesthesiology. 2008 Apr;108(4):703-13. doi: 10.1097/ALN.0b013e318167af46. PMID 18362603